CLINICAL TRIAL: NCT03478774
Title: Physiology Regarding Apnoeic Oxygenation During Nasal Cannula Therapy at Different Flow Rates
Acronym: PHARAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-00293
Record Dates: First submitted 2018-03-08; First posted 2018-03-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Apnoeic Oxygenation
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: single centre, prospective, randomized-controlled trial
Who Masked: Participant
Masking Description: Patients will be blinded as they receive general anesthesia. Care providers cannot be blinded, due to obvious differences in set-up of the different interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (Active Comparator): These patients will receive HFNCT with oxygen 70l/min after induction of general anesthesia. Throughout the entire measurement period of 15 or 30 minutes, continuous videolaryngoscopy will be performed.
  Interventions: Drug: Oxygen 70l/min; Procedure: Videolaryngoscopy
- High flow (Experimental): These patients will receive HFNCT with oxygen 70l/min after induction of general anesthesia. Throughout the entire measurement period of 15 or 30 minutes, jaw thrust will be performed.
  Interventions: Drug: Oxygen 70l/min; Procedure: Jaw thrust
- medium flow (Experimental): These patients will receive oxygen 10l/min after induction of general anesthesia. Throughout the entire measurement period of 15 or 30 minutes, jaw thrust will be performed.
  Interventions: Drug: Oxygen 10 l/min; Procedure: Jaw thrust
- low flow (Experimental): These patients will receive oxygen 2l/min after induction of general anesthesia. Throughout the entire measurement period of 15 or 30 minutes, jaw thrust will be performed.
  Interventions: Drug: Oxygen 2l/min; Procedure: Jaw thrust
- minimal flow (Experimental): These patients will receive a standard tracheal tubes after induction of general anesthesia, with 100% Oxygen and Minimum-flow 0.25l/min. The measurement period is 15 or 30 minutes.
  Interventions: Drug: oxygen 0.25l/min

INTERVENTIONS:
Drug: Oxygen 70l/min — HFNCT will be provided using OptiFlow by Fisher&Paykel.
  Other Names: high flow
  Arms: Control; High flow
Drug: Oxygen 10 l/min — Medium flow will be applied with a humidifier (Hudson RCI) and a standard nasal cannula.
  Other Names: medium flow
  Arms: medium flow
Drug: Oxygen 2l/min — Low flow will be applied with a humidifier (Hudson RCI) and a standard nasal cannula.
  Other Names: low flow
  Arms: low flow
Procedure: Jaw thrust — Continuous
  Arms: High flow; low flow; medium flow
Procedure: Videolaryngoscopy — Continuous
  Arms: Control
Drug: oxygen 0.25l/min — 0.25l/min of oxygen via an endotracheal tube
  Other Names: minimal flow
  Arms: minimal flow

SUMMARY:
This study compares under controlled conditions if different flow rates affect apnoea time after induction of anaesthesia and how CO2 clearance is influenced. Furthermore, this study enables to quantify the effects of increased pCO2 on vital parameters (e.g. blood pressure, cardiac output, cerebral perfusion, etc.) The investigators will enroll patients undergoing elective surgery at the University Hospital of Bern, Switzerland.

Once anesthesia has been induced, apnoea will set it. During this period, the investigators will compare different methods of apnoeic oxygenation for a maximum of 15 or 30 minutes.

Before discharge, an interview will be conducted, assessing complications and patient satisfaction.

DETAILED DESCRIPTION:
Eligible, consenting adults will be prepared for general anaesthesia in the usual way consisting of ECG, pulse-oximetry, NarcotrendTM, a venous cannula and an arterial line for continuous blood pressure monitoring. They will receive additional monitoring such as transcutaneous measurement of pCO2 and O2, NIRS, and thoracic electrical impedance tomography (EIT, PulmoVista® 500, Draeger, Luebeck, Germany).

Normal pre-oxygenation (until etO2 is > 90% or time > 3 minutes) will occur. Anaesthesia will be started (= "induction") using Propofol and Fentanyl, using NarcotrendTM to measure depth of anaesthesia. All patients will receive a standard dose of neuromuscular blockage to facilitate airway management and total intravenous anaesthesia will be installed. Using the train of four measurement (TOF) full neuromuscular blockage with Rocuronium will be confirmed every 30 seconds. If necessary, additional dosage of neuromuscular blockage will be administered.

After administration of Rocuronium, possibility of mask ventilation will be confirmed and the sealed envelope with the randomization will then be opened. As a study intervention, the assigned method (HFNCT 70 l/min with either jaw thrust or laryngoscopy, or 10 l/min or 2l/min with the standard nasal canula, or 0.25l/min delivery of oxgen via a tracheal tube) will be installed and mask ventilation discontinued starting the apnoea period. Nasopharyngoscopy (EF-N slim, Acutronic, Hirzel, Switzerland) will confirm upper airway patency. Blood gas analysis will be conducted: baseline awake, start of apnoea, first minute after apnoea start, and every 2 minutes thereafter with a maximum of 75ml 150 ml in total. Other measurements (ECG, pulse-oximetry, blood pressure, NIRS, thoracic EIT, NarcotrendTM, PtcO2, PtcCO2) will be measured continuously over the study period The study intervention will end when one of the following criteria (study end-points) is met: SpO2 <92%, PtcCO2 > 100 mmHg or time > 30 minutes.

When any of the end points is reached, patient-centred standard anaesthesia care will be continued, as planned for the case.

A post-operative interview will be conducted before discharge to evaluate injuries during airway management (bleeding, sore throat, hoarseness), pain, postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Written informed consent
* Undergoing elective surgery
* Requiring general anesthesia

Exclusion Criteria:

* Any Indication for fibre optic intubation
* Expected impossible mask ventilation
* Known coronary heart disease
* Known heart failure, NYHA classification ≥ 2
* Therapy including β-receptor antagonists
* Arrhythmias in need of anti-arrhythmic therapy (e.g. implanted cardio defibrillator)
* Peripheral occlusive arterial disease, Fontaine ≥ 2b
* Known stenosis of the (common or internal) carotid or vertebral arteries
* BMI > 35kg/m2 and BMI < 16kg/m2
* Hyperkalaemia (K > 5.5 mmol/l)
* Known COPD Gold classification ≥ 2
* Known pulmonary arterial hypertension, systolic > 35mmHg
* Known obstructive sleep apnoea syndrome in need of therapy
* High risk of aspiration (requiring rapid sequence induction intubation)
* Increased intracranial pressure
* Intracranial surgery
* Limited knowledge of German language
* Absent power of judgement
* Anaemia, Hb < 100 g/l
* Pregnancy (pregnancy test in all female patients)
* Neuromuscular disorder
* Known or suspected cervical spine instability
* Nasal obstruction, impossibility of nasal ventilation (both sides patent)
* Allergies or contra-indications to one or more of the used anaesthesia agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
pCO2 increase in kPa/min | 15 or 30 minutes (maximum apnea time)
  pCO2 will be measured transcutaneously throughout the apnea period

SECONDARY OUTCOMES:
Lowest Saturation | During apnea period (until end-point is met or max. 15 or 30 minutes)
  Lowest SpO2 in %
Change in PaO2 in kPa | During apnea period (until end-point is met or max. 15 or 30 minutes)
  Blood gas analyses as well as transcutaneous measurement
Change in cardiac output in L/min | During apnea period (until end-point is met or max. 15 or 30 minutes)
  Cardiac output will be measured using pulse pressure measurement
Change in cerebral perfusion in % | During apnea period (until end-point is met or max. 15 or 30 minutes)
  Near infrared spectroscopy will be measured continuously
Changes in end-expiratory lung impedance | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  To quantify atelectasis during apnoeic oxygenation
Change in invasive blood pressure | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  Measurement of change due to hypercarbia
Standard monitoring | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  3 pole ECG
Depth of anaesthesia | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  Using Narcotrend-EEG
Bilateral brain oxygenation | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  Using NIRS
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  pH
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  pCO2 in mmhg
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  pO2 in mmhg
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  SaO2 in %
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  Potassium in mmol
Arterial blood gas analyses | At 0, 1, 3, 5, 7, 9, 11, 13 and 15 minutes of apnoea or 0,1,3,5,7,9,13,15,17,19,21,23,25,27,29 and 30 min of apnoea.
  Bicarbonate in mmol
Postoperative questionnaire | Morning of first postoperative day
  Visual analogue scale (VAS) : pain, nausea, vomiting, feeling worried or anxious, feeling sad or depressed, injuries, discomfort, any complications
Standard monitoring | During apnoea time (until end-point is met or max. 15 or 30 minutes)
  Pulse oximetry SpO2 in %

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Theiler, PD MD, Principal Investigator — University hospital of Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407
- [Derived] Schweizer T, Hartwich V, Riva T, Kaiser H, Theiler L, Greif R, Nabecker S. Limitations of transcutaneous carbon dioxide monitoring in apneic oxygenation. PLoS One. 2023 Jun 1;18(6):e0286038. doi: 10.1371/journal.pone.0286038. eCollection 2023. PMID 37262066
- [Derived] Riedel T, Burgi F, Greif R, Kaiser H, Riva T, Theiler L, Nabecker S. Changes in lung volume estimated by electrical impedance tomography during apnea and high-flow nasal oxygenation: A single-center randomized controlled trial. PLoS One. 2022 Sep 28;17(9):e0273120. doi: 10.1371/journal.pone.0273120. eCollection 2022. PMID 36170281
- [Derived] Theiler L, Schneeberg F, Riedel T, Kaiser H, Riva T, Greif R. Apnoeic oxygenation with nasal cannula oxygen at different flow rates in anaesthetised patients: a study protocol for a non-inferiority randomised controlled trial. BMJ Open. 2019 Jul 11;9(7):e025442. doi: 10.1136/bmjopen-2018-025442. PMID 31300494